CLINICAL TRIAL: NCT04098432
Title: Stereotactic Radiotherapy + Anti PD-1 Therapy in Patients with Locally Advanced Unresectable Pancreatic Adenocarcinoma
Brief Title: STR + Anti PD-1 Therapy in Patients with Locally Advanced Unresectable Pancreatic Adenocarcinoma
Acronym: CA209-9KH
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Hospital Hradec Kralove (Other)
Collaborators: Bristol-Myers Squibb (Industry); GCP-Service International s.r.o. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA209- 9KH
Record Dates: First submitted 2019-03-06; First posted 2019-09-23 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Locally Advanced Unresectable Pancreatic Adenocarcinoma
Keywords: Stereotactic radiotherapy; Nivolumab; Anti PD-1; Pancreatic cancer; Pancreatic Adenocarcinoma
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Nivolumab; Radiosurgery; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Arm 1 (Experimental): 4-weeks stereotactic radiotherapy followed by nivolumab 3 mg/kg every two weeks
  Interventions: Drug: Nivolumab; Radiation: Stereotactic radiotherapy

INTERVENTIONS:
Drug: Nivolumab — Nivolumab 3 mg/kg intravenously every two weeks untill disease progression or unacceptable toxicity
  Other Names: Opdivo
Radiation: Stereotactic radiotherapy — The prescribed dose will be 32 Gy in four fractions in four weeks (8 Gy per one fraction).
  Other Names: Radiation

SUMMARY:
Stereotactic Radiotherapy + Anti PD-1 Therapy in Patients With Locally Advanced Unresectable Pancreatic Adenocarcinoma

DETAILED DESCRIPTION:
Phase I/II, multicentre, open label, with no control arm clinical trial of 4-weeks stereotactic radiotherapy followed by nivolumab 3 mg/kg every two weeks in adults with locally advanced pancreatic cancer who does not progress during 4 cycles of standard chemotherapy FOLFIRINOX

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients aged ≥18 years
2. Eastern Cooperative Oncology Group (ECOG) performance score of 0 or 1
3. Locally advanced, unresectable, histologically confirmed primary adenocarcinoma of pancreas with no progression during induction chemotherapy (4 cycles of FOLFIRINOX - not a part of trial). Within screening period tumor tissue must be available and sent to the central pathological reviewer in order to confirm the diagnosis.
4. Measurable (one target lesion is sufficient) disease as per RECIST 1.1 criteria
5. Laboratory values:

   1. Aspartate aminotransferase (AST) ≤ 3x ULN (upper limit of normal)
   2. Alanine transaminase (ALT) ≤ 3x ULN
   3. Total bilirubin ≤ 1.5 x ULN (except subjects with Gilbert syndrome who must have a total bilirubin ≤ 3x ULN)
   4. Creatinine: Serum creatinine ≤ 1.5 ULN or creatinine clearance > 50ml/min (using Cockcroft/Gault formula)
   5. White blood cells ≥ 2000 /ul
   6. Neutrophils ≥ 1500 /ul
   7. Platelets ≥ 100x 103 /ul
   8. Hemoglobin ≥ 9.0 g/l
6. Women of childbearing potential (WOCBP) must have a negative serum pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 24 hours prior to the start of study treatment. WOCBP is defined as any female who has experienced menarche and who has not undergone surgical sterilization (hysterectomy or bilateral oophorectomy) and who is not postmenopausal. Menopause is defined as 12 months of amenorrhea in a woman over age 45 years in the absence of other biological or physiological causes. In addition, females under age of 55 years must have serum follicle stimulating hormone (FSH) level > 40mIU/ml to confirm menopause.

Exclusion Criteria:

1. Other histology then primary pancreatic adenocarcinoma
2. Resectable disease
3. Distant metastases
4. Progressive disease during induction chemotherapy (4 cycles of FOLFIRINOX)
5. Other previous treatment of the disease except induction chemotherapy (4 cycles of FOLFIRINOX)
6. ECOG performance score of 2 or more
7. Previous therapy of malignant disease in 5 years and less before inclusion to the trial (except skin epithelial tumors)
8. Previous radiotherapy in abdominal region
9. Previous immunological treatment (anti-CTLA-4, anti-PD1 or anti-PD-L1)
10. Active, known or suspected serious autoimmune disease
11. Major surgery less than 28 days prior to the first dose of study treatment
12. Treatment of any investigational medicinal product within 4 weeks before this trial enrolment
13. Any positive test for hepatitis B virus or hepatitis C virus indicating acute or chronic infection
14. Known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency synrome (AIDS)
15. Prisoners or subjects who are involuntarily incarcerated
16. Subjects who are compulsorily detained for treatment of either a psychiatric or physical (e.g. infectious disease) illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2018-12-03 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Safety - incidence of treatment-related adverse events | Through study completion, an average of 4 years
  Measured by the incidence of adverse events (AEs), serious adverse events (SAEs), deaths
Safety - incidence of laboratory abnormalities | Through study completion, an average of 4 years
  Biochemistry - Na (mmol/l), K (mmol/l), Cl (mmol/l), Ca (mmol/l), Ca ionized (mmol/l), Mg (mmol/l), P (mmol/l), urea (mmol/l), creatinine (µmol/l), LDH (µkat/l), AST(µkat/l), ALT(µkat/l), ALP(µkat/l), GMT(µkat/l), total bilirubin (µmol/l), conjuged bilirubin (µmol/l), total protein (g/l), albumin (g/l), fasting glucose (mmol/l), amylase (µkat/l), C-reactive protein (mg/l), endocrine panel - TSH (mU/l), Free T3 (pmol/l), Free T4 (pmol/l), hematology - complete blood count (CBC): hemoglobin (g/l), hematocrit (ratio), white blood cells (WBC) (10E9/l), red blood cells (10E12/l), platelets (10E9/l) including differential (all 10E9/l), coagulation - APTT (ratio), PT (ratio)

SECONDARY OUTCOMES:
Progression free survival | Through study completion, an average of 4 years
  To evaluate progression free survival (median of progression free survival and 1-, 2-year progression free survival)
Overall survival | Through study completion, an average of 4 years
  To evaluate overall survival (median of overall survival and 1-, 2-year overall survival)
Relationship of laboratory markers and progression | Through study completion, an average of 4 years
  To evaluate the relationship of laboratory markers (PD-L1 expression, tumor infiltrating lymphocytes presence, neopterin level) to progression status and time related progress of biomarkers (CEA, CA19-9)
patient's capacity to fulfill the activities of daily living and quality of life | Through study completion, an average of 4 years
  Assess by questionnaire European Organisation for Research and Treatment of Cancer (EORTC) Quality of life questionnaire (QLQ-C30) questionnaire. The EORTC QLQ-C30 comprises 30 items (i.e. single questions), 24 of which are aggregated into 9 multi-item scales, that is, 5 functioning scales (physical, role, cognitive, emotional and social), 3 symptom scales (fatigue, pain and nausea/vomiting) and one global health status scale. The remaining 6 single-item (dyspnoea, appetite loss, sleep disturbance, constipation, diarrhoea and the financial impact) scales assess symptoms.All of the scales and single-item measures range in score from 0 to 100. Higher score for the functioning scales and global health status denote a better level of functioning (i.e. a better state of the patient), while higher scores on the symptom and single-item scales indicate a higher level of symptoms (i.e. a worse state of the patient).

CONTACTS AND LOCATIONS:
Locations (4):
- Czechia (4):
  - Klinika Onkologie a radioterapie, Fakultní nemocnice Hradec Králové, Hradec Králové
  - Onkologická klinika, Fakultní nemocnice Olomouc, Olomouc
  - Onkologická klinika, Thomayerova nemocnice, Prague
  - Ústav radiační onkologie, Nemocnice Na Bulovce, Prague

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vosmik M, John S, Dvorak J, Mohelnikova-Duchonova B, Melichar B, Lohynska R, Ryska A, Banni AM, Krempova J, Sirak I. Stereotactic Radiotherapy Plus Nivolumab in Patients with Locally Advanced Pancreatic Cancer: Results from Phase 1/2 Clinical CA209-9KH Trial. Oncol Ther. 2024 Dec;12(4):817-831. doi: 10.1007/s40487-024-00309-z. Epub 2024 Oct 23. PMID 39441483